CLINICAL TRIAL: NCT04848506
Title: A Follow-Up, Open-Label, Research Evaluation of Sustained Treatment With Aficamten (CK-3773274) in Hypertrophic Cardiomyopathy (HCM)
Brief Title: Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of Aficamten in Adults With HCM
Acronym: FOREST-HCM
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CY 6022; 2020-003571-17 (EudraCT Number); 2023-508963-58-00 (Other: EU CTR Number)
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Symptomatic Hypertrophic Cardiomyopathy (HCM)
Keywords: Obstructive Hypertrophic Cardiomyopathy; oHCM; CK-3773274; CK-274; Non obstructive hypertrophic cardiomyopathy; nHCM; HCM; Hypertrophic cardiomyopathy; Aficamten; REDWOOD-OLE; CY 6022; FOREST-HCM; Forest
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aficamten up to 20 mg (Experimental): Patients in this arm take daily dose of aficamten. Each patient will start at the lowest prespecified dose and titrate up to their maximum tolerated dose.
  Interventions: Drug: Aficamten (5 - 20 mg)

INTERVENTIONS:
Drug: Aficamten (5 - 20 mg) — Aficamten tablets administered orally. During titration phase, clinic visits will occur approximately every 2-6 weeks. In the maintenance phase clinic visits will occur every 24 weeks, with safety check-in occurring every 12 weeks between visits by phone or, if desirable, in the clinic.

SUMMARY:
The purpose of this study is to collect long-term safety and tolerability data for aficamten.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a Cytokinetics trial investigating aficamten
* LVEF ≥ 55% at the Screening Visit

Exclusion Criteria:

* Has received treatment with mavacamten: (a) within 56 days prior to dosing and (b) has not received approval for participation from the Medical Monitor.
* Has participated in another investigational device or drug study or received an investigational device or drug < 1 month (or 5 half-lives for drugs, whichever is longer) prior to screening. Other investigational procedures while participating in this study are not permitted.
* Since completion of a previous trial of aficamten has:

  * Developed new-onset paroxysmal or permanent atrial fibrillation requiring rhythm restoring treatment (eg, direct-current cardioversion, ablation procedure, or antiarrhythmic therapy) < 30 days prior to screening. Patient may re-screen for CY 6022 after 30 days if heart rate (HR) < 100 bpm and/or rhythm is stable > 30 days
  * Undergone septal reduction therapy (surgical myectomy or transcatheter alcohol ablation)
* Had a confirmed LVEF < 40% with an associated dose interruption during participation in a prior study with aficamten
* History of implantable ICD placement within 30 days prior to screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events observed during dosing of aficamten in patients with HCM | Baseline to End of study, up to 5 years
  Patient incidence of reported Adverse Events (AEs)

SECONDARY OUTCOMES:
Incidence of serious adverse events observed during dosing of aficamten in patients with HCM | Baseline to End of study, up to 5 years
  Patient incidence of reported Serious Adverse Events (SAEs)
Incidence of left ventricular ejection fraction (LVEF) < 50% observed during dosing of aficamten in patients with HCM | Baseline to End of study, up to 5 years
  Patient incidence of reported LVEF <50%
Long-term effects of aficamten on left ventricular outflow tract gradient (LVOT G) in patients with oHCM | Baseline through the end of participation at 12-24 week intervals
  Peak LVOT-G at rest; applicable only to patients with oHCM
Long-term effects of aficamten on resting LVOT-G | Baseline through the end of participation at 12-24 week intervals
  Proportion of patients with resting LVOT-G < 30 mmHg; applicable only to patients with oHCM
Long-term effects of aficamten on post Valsalva LVOT-G | Baseline through the end of participation at 12-24 week intervals
  Proportion of patients with post-Valsalva LVOT-G < 50 mmHg; applicable only to patients with oHCM
Long-term effects of aficamten on post Valsalva LVOT-G | Baseline through the end of participation at 12-24 week intervals
  Proportion of patients with post-Valsalva LVOT-G < 30 mmHg; applicable only to patients with oHCM
Long-term effects of aficamten on left ventricular ejection fraction (LVEF) and post-Valsalva LVOT-G | Baseline through the end of participation at 12-24 week intervals
  Proportion of patients with LVEF ≥ 50%, resting LVOT-G < 30 mmHg, and post-Valsalva LVOT-G < 50 mmHg; applicable only to patients with oHCM
Long-term effects of aficamten on time to first resting LVOT-G < 30 mmHg through last follow-up | Time to the following event through last follow-up, up to 5 years
  Applicable only to patients with oHCM
Long-term effects of aficamten on time to first post-Valsalva LVOT-G < 50 mmHg through last follow-up | Time to the following event through last follow-up, up to 5 years
  Applicable only to patients with oHCM
Long-term effects of aficamten on time to first post-Valsalva LVOT-G < 30 mmHg through last follow-up | Time to the following event through last follow-up, up to 5 years
  Applicable only to patients with oHCM
Long-term effects of aficamten on time to first LVEF ≥ 50%, resting LVOT-G < 30 mmHg, and post-Valsalva LVOT-G < 50 mmHg through last follow-up | Time to the following event through last follow-up, up to 5 years
  Applicable only to patients with oHCM

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics, MD, Study Director — Cytokinetics
Locations (129):
- United States (52):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alaska Heart and Vascular Institute, Anchorage, Alaska
  - Mayo Clinic Building - Phoenix, Phoenix, Arizona
  - UC San Diego Health - Sulpizio Cardiovascular Center, La Jolla, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center (Smidt Heart Institute), Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital / Cardiology Associates, Fort Lauderdale, Florida
  - Emory Clinic, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northwestern University, Evanston, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Michigan Medicine - University of Michigan, Ann Arbor, Michigan
  - University of Michigan Health System (UMHS) - University Hospital (University of Michigan Medical Center), Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Northwell Health North Shore University Hospital, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Sanger Heart & Vascular Institute - HCM Clinic, Charlotte, North Carolina
  - Duke Cardiology at Southpoint, Durham, North Carolina
  - The Linder Research Center at The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania (University of Pennsylvania School of Medicine), Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Ascension Saint Thomas Heart West, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia Health System University Hospital, Charlottesville, Virginia
  - Inova Health Care Services, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - WVUMedicine, Morgantown, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Instituto Cardiovascular de Buenos Aires(ICBA), Buenos Aires, Argentina
- Australia (3):
  - Flinders Medical Centre, Cardiology Research, Bedford Park
  - The Prince Charles Hospital, Chermside
  - Fiona Stanley Hospital, AHF Unit, Murdoch
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Canada (3):
  - Institut universitaire de cardiologie et de pneumologie de Quebec-Universite Laval, Québec, Quebec
  - Royal Alexandra Hospital, Edmonton
  - QEII Health Science Centre (Halifax Infirmary site), Halifax
- Il. Interni klinika kardiologie a angiologie, Prague, Czechia
- Denmark (5):
  - Department of Cardiology Aalborg University Hospital, Aalborg
  - Department of Cardiology Aarhus University Hospital, Aarhus
  - The Heart Center, Department of Cardiology, Copenhagen
  - Copenhagen University Hospital, Copenhagen
  - Odense University Hospital, Odense
- France (9):
  - Hopital de la Timone Service de cardiologie, Marseille
  - Clinique Du Millenaire, Montpellier
  - CHU Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - CHU de Nantes Institut Du Thorax et du systeme nerveux Clinique Cardiologique et des Maladies Vasculaires, Nantes
  - Hopital Lariboisiere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital cardiologique de Haut-Leveque, Pessac
  - Centre hospitalier universitaire (CHU) de Rennes-Hopital Pontchaillou, Rennes
  - Centre Hospitalier universitaire de Toulouse - Rangueil Hospital, Toulouse
- Germany (6):
  - Charite-Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsmedizin Goettingen Klinik fur Kardiologie und Pneumologie, Goettigen
  - Universitaesklinkum Heidelberg, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetskinikum Wuerzburg Deutsches Zentrum fur Herzinsuffzienz Wurzburg (DZHI) Comprehensive Heart Failure Center (CHFC), Würzburg
- Greece (4):
  - Evangelismos General Hospital of Athens, Athens
  - "Hippokration" General Hospital of Athens, Athens
  - Onassis Hospital, Athens
  - University General Hospital "ATTIKON", Attiki
- Hungary (2):
  - Semmelweis Egyetem Varosmajori Sziv es Ergyogyaszati Klinika, Budapest
  - Szegedi Tudományegyetem, Belgyógyászati Klinika, Kardiológiai Központ, Szeged
- Landspitali University Hospital, Reykjavik, Iceland
- Israel (5):
  - The Barzilai University Medical Center, Ashkelon
  - Hadassah Medical Center- Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center, Ramat Gan
  - Ziv Medical Center, Safed
- Italy (7):
  - Unit Cardiomiopatie, Dipartimento Cardio ToracoVascolare, Florence
  - IRCCS Policlinico San Donato, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - Fondazione toscana Gabriele Monesterio per la ricarca medica Dipartimento Cardiotoracico UOC Cardiologia e Medicina Cardiovasculare Ospedale San Cataldo, Pisa
  - Dipartimento di Medicina Clinica e Molecolare Universita Sapienza di Roma Unita di Terapia Intensiva Cardiologica Azienda Ospedaliero Universitaria Sant'Andrea, Roma
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Maastricht University Medical Center (MUMC), Maastricht
  - Erasmus Medical Center Department of Cardiology, Rotterdam
- Poland (2):
  - Kardio Brynow S.C., Katowice
  - Narodowy Instytut Kardiologii Stefana Kardynala Wyszynskiego - Panstwowy Instytut Badawczy Centrum Zaburzen Rytmu Serca, Warsaw
- Portugal (4):
  - Centro Hospitalar Do Baixo Vouga, EPE Cardiology Department, Aveiro
  - Unidade Local De Saude De Sao Jose E.P.E, Lisbon
  - Hospital Cuf Descobertas S.A., Lisbon
  - Hospital da Luz, Lisbon
- Spain (12):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón (HGUGM), Madrid
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Son Llatzer, Palma
  - Complexo Hospitalario Universitario De Vigo, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena-merge, Seville
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Ninewells Hospital and Medical School, Dundee
  - Glasgow Clinical Research Facility Neuroscience Institute, Glasgow
  - Liverpool Heart and Chest Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Royal Brompton Hospital, London
  - Oxford Centre for Clinical Magnetic Resonance Research (OCMR) Division of Cardiovascular Medicine Radcliffe Department of Medicine University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saberi S, Abraham TP, Choudhury L, Barriales-Villa R, Elliott PM, Nassif ME, Oreziak A, Owens AT, Tower-Rader A, Rader F, Garcia-Pavia P, Olivotto I, Coats CJ, Fifer MA, Sherrid MV, Solomon SD, Watkins H, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Melloni C, Meng L, Wei J, Maron MS, Masri A; FOREST-HCM Steering Committee and Investigators. Aficamten Treatment for Symptomatic Obstructive Hypertrophic Cardiomyopathy: 48-Week Results From FOREST-HCM. JACC Heart Fail. 2025 Aug;13(8):102496. doi: 10.1016/j.jchf.2025.03.040. Epub 2025 Jun 19. PMID 40540987
- [Derived] Masri A, Maron MS, Abraham TP, Nassif ME, Barriales-Villa R, Bilen O, Coats CJ, Elliott P, Garcia-Pavia P, Massera D, Olivotto I, Oreziak A, Owens AT, Saberi S, Solomon SD, Tower-Rader A, Heitner SB, Jacoby DL, Melloni C, Wei J, Sherrid MV; REDWOOD-HCM, SEQUOIA-HCM, and FOREST-HCM Investigators. Concomitant Aficamten and Disopyramide in Symptomatic Obstructive Hypertrophic Cardiomyopathy. JACC Heart Fail. 2025 Apr 2:102441. doi: 10.1016/j.jchf.2025.03.008. Online ahead of print. PMID 40285763
- [Derived] Masri A, Choudhury L, Barriales-Villa R, Elliott P, Maron MS, Nassif ME, Oreziak A, Owens AT, Saberi S, Tower-Rader A, Rader F, Garcia-Pavia P, Olivotto I, Nagueh SF, Wang A, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Melloni C, Meng L, Wei J, Sherrid MV, Abraham TP; FOREST-HCM Investigators. Standard-of-Care Medication Withdrawal in Patients With Obstructive Hypertrophic Cardiomyopathy Receiving Aficamten in FOREST-HCM. J Am Coll Cardiol. 2024 Nov 5;84(19):1839-1849. doi: 10.1016/j.jacc.2024.09.002. PMID 39477631